CLINICAL TRIAL: NCT04882072
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study of Ustekinumab in Participants With Takayasu Arteritis
Brief Title: A Study of Ustekinumab in Participants With Takayasu Arteritis (TAK)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to difficulties in enrollment and ongoing feasibility issues
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108981; CNTO1275TAT3001 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2021-05-10; First posted 2021-05-11 (Actual); Results first posted 2024-12-02 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Takayasu Arteritis
MeSH Terms: conditions — Takayasu Arteritis | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ustekinumab (Experimental): Double-blind (DB) Period: Participants will receive weight-ranged based ustekinumab (6 milligrams/kilogram[mg/kg]) as IV infusion at Week 0 followed by ustekinumab 90mg injection SC 8 weeks after initial IV dose, then every 8 weeks (q8w) thereafter until the end of the DB period with starting the protocol defined oral GC taper regimen from Week 2 visit.
  Open Label Extension (OLE) period: Participants will receive ustekinumab SC injection at Week OL-0, followed by ustekinumab 90mg SC injection with oral GC taper at investigator's discretion for 52 weeks (Week OL-52) or until 32 weeks from first SC administration after end of DB period whichever is later.
  Long-term Extension (LTE) Period: Participants who completed OLE period may be eligible to enter LTE and continue to receive ustekinumab 90mg SC injection q8w.
  Interventions: Drug: Ustekinumab; Drug: Glucorticoid Taper Regimen
- Placebo (Placebo Comparator): DB period: Participants will receive placebo intravenous (IV) infusion at Week 0 followed by placebo subcutaneous (SC) injection administration, 8 weeks after the initial IV dose, then q8w thereafter until the end of DB period with starting the protocol defined oral GC taper regimen from Week 2 visit.
  OLE period: Participants will receive ustekinumab SC at Week OL-0, followed by SC administration of ustekinumab with oral GC taper at investigator's discretion for 52 weeks (Week OL-52) or until 32 weeks from the first SC administration after the end of DB period, whichever is later.
  LTE Period: Participants who complete their participation in OLE period may be eligible to enter the LTE and continue to receive 90 mg SC ustekinumab q8w.
  Interventions: Drug: Ustekinumab; Other: Placebo; Drug: Glucorticoid Taper Regimen

INTERVENTIONS:
Drug: Ustekinumab — Participants will receive IV infusion and SC injection of ustekinumab.
  Other Names: Stelara®; CNTO1275
Other: Placebo — Participants will receive IV infusion and SC injection of matching placebo.
  Arms: Placebo
Drug: Glucorticoid Taper Regimen — Glucocorticoid will be administered orally.

SUMMARY:
The purpose of this study is to evaluate the efficacy of ustekinumab compared to placebo, in combination with oral glucocorticoid (GC) taper regimen, in participants with relapsing Takayasu Arteritis (TAK).

ELIGIBILITY:
Inclusion Criteria:

* Must have developed a relapse of Takayasu Arteritis (TAK) within 12 weeks prior to administration of study intervention and the relapse must have occurred at a dose of at least 7.5 milligrams (mg)/day (prednisolone or equivalent)
* Must be receiving oral glucorticoid (GC) treatment of greater than or equal to (>=)15 mg/day (prednisolone or equivalent), inclusive for the treatment of relapsing TAK and be on a stable dose for at least 2 weeks prior to the first administration of study intervention
* If receiving an oral anti-platelet therapy (including but not limited to aspirin, clopidogrel, ticlopidine) or anti-coagulation therapy (including but not limited to warfarin) for treatment of TAK, the dose must have been stable for at least 2 weeks prior to first administration of the study intervention. In terms of warfarin, the dose should be controlled 1-5mg/day to maintain Prothrombin Time and International Normalized Ratio (PT-INR) target range between 2.0-3.0 (if participants are over 70 years old, PT-INR target range should be between 1.6-2.6)
* Have no history of latent or active Tuberculosis (TB) prior to screening. An exception is made for participants who have a history of latent TB and are currently receiving treatment for latent TB, will initiate treatment for latent TB at least 3 weeks prior to the first administration of the study intervention, or have documentation of having completed appropriate treatment for latent TB within 3 years prior to the first administration of the study intervention. It is the responsibility of the investigator to verify the adequacy of previous antituberculous treatment and provide appropriate documentation
* If receiving an oral anti-hypertensive therapy for treatment of TAK, the dose must have been stable for at least 2 weeks prior to first administration of the study intervention

Exclusion Criteria:

* Has currently any known severe or uncontrolled TAK complications (example, hypertension not responding to adequate treatment, aortic incompetence with cardiac insufficiency, progressing aortic aneurysm, coronary artery lesions with severe stenosis)
* Has received immunosuppressant (s) (including but not limited to Methotrexate [MTX], Azathioprine [AZA], Mycophenolate Mofetil [MMF], oral Triamcinolone [TAC], oral Cyclosporine A) within 4 weeks of first study intervention
* Has had a Bacille Calmette-guerin (BCG) vaccination within 12 months of screening
* Any major illness/condition or evidence of an unstable clinical condition example, history of liver or renal insufficiency (estimated creatinine clearance below 60 milliliters/minute [mL/min]); significant (cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances), disease of any organ system or active acute or chronic infection/infectious illness that, in the investigator's judgment, will substantially increase the risk to the participant if he or she participates in the study
* Having a condition that is steroid dependent (example, steroid dependent asthma, chronic obstructive pulmonary disease, et cetera) that is not amenable to tapering oral GC

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (27):
- Japan (27):
  - Tokyo Medical and Dental University Hospital, Bunkyō City
  - Chiba University Hospital, Chiba
  - Kyushu University Hospital, Fukuoka
  - Hamamatsu University Hospital, Hamamatsu
  - Saitama Medical University Hospital, Iruma-gun
  - Kagawa University Hospital, Kita Gun
  - Kobe University Hospital, Kobe
  - Kyoto University Hospital, Kyoto
  - Matsuyama Red Cross Hospital, Matsuyama
  - Nagoya City University Hospital, Nagoya
  - Niigata University Medical And Dental Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Kitano Hospital, Osaka
  - Rinku General Medical Center, Osaka
  - Kindai University Hospital, Osaka Sayama Shi
  - Kitasato University Hospital, Sagamihara
  - Sapporo Medical University Hospital, Sapporo
  - Hokkaido University Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku Ku
  - National Cerebral and Cardiovascular Center, Suita-Shi
  - Mitsui Memorial Hospital, Tokyo
  - St. Luke's International Hospital, Tokyo
  - Fujita Health University Hospital, Toyoake
  - University of Tsukuba Hospital, Tsukuba
  - Wakayama Medical University Hospital, Wakayama
  - Tottori University Hospital, Yonago

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Yoshifuji H, Ishii T, Ohashi H, Yoshizawa K, Mihoya M, Nishikawa K, Nakaoka Y. Phase 3, multicentre, randomized, double-blind, placebo-controlled, parallel-group study of ustekinumab in patients with Takayasu arteritis. Rheumatol Adv Pract. 2025 Feb 3;9(2):rkaf013. doi: 10.1093/rap/rkaf013. eCollection 2025. PMID 40104212

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to the early study termination, participants who had relapse during double blind period were only able to enter open label extension (OLE) period.
Groups:
- Placebo Then Ustekinumab: In the double blind-period, participants received placebo matched to ustekinumab as intravenous (IV) infusion at Week 0 followed by placebo subcutaneous (SC) injection at Week 8 and thereafter every 8 weeks (q8w) until developing relapse or end of double blind period (up to 8.1 weeks), with starting the protocol defined oral glucocorticoid (GC) taper regimen from Week 2. Upon relapse, participants received rescue medication of greater than or equal to (>=) doubled oral GC dose. These participants were assessed whether they achieved remission at the next scheduled dose administration visit (open label [OL] Week 0) from the relapse to enter OLE period and then they received ustekinumab 90 mg IV infusion at OL Week 0 followed by ustekinumab 90 mg SC injection at OL Week 8 and thereafter q8w in OLE period (maximum exposure: 48.1 weeks). Rest of the participants entered OLE period after end of double blind-period and received ustekinumab 90 mg SC injection (maintenance dosing) q8w from OL Week 0 (maximum exposure: 48.1 weeks). Participants who reached oral GC dose of 5 mg/day or less at the end of double blind period were terminated from study intervention administration and underwent early-term visit after completion of double blind period.
- Ustekinumab Then Ustekinumab: In the double-blind period, participants received body weight-range based ustekinumab (6 mg/kg) IV infusion at Week 0 followed by ustekinumab 90 mg SC injection at Week 8 and thereafter q8w until developing relapse or end of double-blind period (maximum exposure: 56.1 weeks), with starting the protocol defined oral GC taper regimen from Week 2. Upon relapse, participants received rescue medication of >=doubled oral GC dose. These participants were assessed whether they achieved remission at the next scheduled dose administration visit (OL Week 0) from the relapse to enter OLE period and then they received ustekinumab 90 mg IV infusion at OL Week 0 followed by ustekinumab 90 mg SC injection at OL Week 8 and thereafter q8w in OLE period (maximum exposure: 48.1 weeks). Rest of the participants entered OLE period after end of double-blind period and received ustekinumab 90 mg SC injection (maintenance dosing) q8w from OL Week 0 (maximum exposure: 48.1 weeks).
Period: Double Blind: Week 0 to Week 71.1
Arm/Group | Placebo Then Ustekinumab | Ustekinumab Then Ustekinumab
Started | 8 | 6
Completed | 6 | 6
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Withdrawal Criterion Met | 1 | 0
Period: OL Extension: OL Week 0 to OL Week 63.1
Arm/Group | Placebo Then Ustekinumab | Ustekinumab Then Ustekinumab
Started | 3 | 4
Completed | 3 | 3
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then Ustekinumab | Ustekinumab Then Ustekinumab | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (15.46) | 36.5 (12.19) | 44 (15.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 6 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse (ToR) of Takayasu Arteritis (TAK) According to Protocol-defined Criteria Through the End of Double-blind Period
Description: ToR:time from randomization to 1st relapse through end of double-blind period (EDBP) per protocol-defined criteria with 5 categories:systemic (objective):body temperature >=38.0°C, weight loss >2kg in 4 weeks, arthralgia, swelling & tenderness =>2 joints; systemic (subjective):malaise, myalgia, headache, dizziness/vertigo at >= grade 2, high inflammation markers (C-reactive protein >=1.0mg/dL, erythrocyte sedimentation rate >=30mm/hr), vascular symptoms:renovascular hypertension: if normal BP <120/80mmHg risen to >=140/90mmHg, or if normal BP >=120/80mmHg, diastolic BP risen by >=20mmHg, new bruits/loss of pulse/difference in systolic BP between left and right by >=10mmHg/tenderness/spontaneous pain in carotid artery/chest/back region, aortic valve incompetence; ischemic symptoms:abdominal pain, seizure, syncope, intermittent claudication, ischemic cardiac pain. Relapse:>=2 categories met criteria.
Time Frame: From double-blind Week 0 up to end of double-blind period (up to 71.1 weeks)
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study intervention through double-blind period. Censored:death/discontinued drugs at last assessment through EDBP (before relapse)/before EDBP (no relapse).
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- Double-blind: Placebo: In double-blind period, participants received placebo matched to ustekinumab as intravenous (IV) infusion at Week 0 followed by placebo subcutaneous (SC) injection administration, 8 weeks after the initial IV dose, then every 8 weeks (q8w) thereafter until developing relapse or end of double-blind period, with starting the protocol defined oral GC taper regimen from Week 2. Participants who received placebo in double-blind period and reached oral GC dose of 5 mg/day or less were terminated from study intervention administration and underwent early-term visit after completion of double-blind period.
- Double-blind: Ustekinumab: Participants received weight-range based ustekinumab (6 milligrams/kilogram [mg/kg]) as IV infusion at Week 0 followed by ustekinumab 90 mg SC injection 8 weeks after initial IV dose, then q8w thereafter until developing relapse or end of double-blind period, with starting the protocol defined oral GC taper regimen from Week 2.
Arm/Group | Double-blind: Placebo | Double-blind: Ustekinumab
Number analyzed (Participants) | 8 | 6
Weeks | 12.64 [12.14 to NA] — Upper limit of 95% confidence interval (CI) was not estimable due to less number of participants with events due to early study termination. | 11.14 [4.14 to NA] — Upper limit of 95% CI was not estimable due to less number of participants with events due to early study termination.
Statistical Analysis 1: Comparison: Double-blind: Placebo vs Double-blind: Ustekinumab; Test type: Superiority; Hazard Ratio (HR) = 1.86, 95% CI 2-sided [0.41 to 8.47]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with the study intervention. TEAEs were defined as AEs with onset or worsening on or after date of first dose of study intervention through the day of last dose.
Time Frame: Double-blind period: Double-blind Week 0 up to end of double-blind treatment period (56.1 weeks); OLE period: OL Week 0 up to end of OLE treatment period (48.1 weeks)
Population: The safety analysis set included all participants who received at least 1 dose of study intervention through double-blind period and OLE period.
Measure: Count of Participants; unit: Participants
Groups:
- OLE: Placebo Then Ustekinumab: Participants who had relapse during the double-blind period, received rescue medication of >=doubled oral GC dose. These participants were assessed whether they achieved remission at the next scheduled dose administration visit (OL Week 0) from the relapse to enter OLE period and received ustekinumab 90 mg IV infusion at OL Week 0 followed by ustekinumab 90 mg SC injection at OL Week 8 and thereafter q8w in OLE period (maximum exposure: 48.1 weeks). Rest of the participants entered OLE period after end of double blind period and then they received ustekinumab 90 mg SC injection (maintenance dosing) q8w from OL Week 0 (maximum exposure: 48.1 weeks). Participants who received placebo (up to 8.1 weeks) in double-blind period received ustekinumab 90 mg SC injection (maintenance dosing) q8w from OL Week 0 till end of OLE period (maximum exposure: 48.1 weeks).
- OLE: Ustekinumab Then Ustekinumab: Participants who had relapse during the double-blind period, received rescue medication of >=doubled oral GC dose. These participants were assessed whether they achieved remission at the next scheduled dose administration visit (OL Week 0) from the relapse to enter OLE period and then they received ustekinumab 90 mg IV infusion at OL Week 0 followed by ustekinumab 90 mg SC injection at OL Week 8 and thereafter q8w till end of OLE period (maximum exposure: 48.1 weeks). Participants with no remission status received ustekinumab IV infusion at OL Week 0 and thereafter q8w till end of OLE period (maximum exposure 48.1 weeks). Rest of the participants entered OLE period after end of double-blind period and received ustekinumab 90 mg SC injection (maintenance dosing) q8w from OL Week 0 (maximum exposure: 48.1 weeks).
Arm/Group | Double-blind: Placebo | Double-blind: Ustekinumab | OLE: Placebo Then Ustekinumab | OLE: Ustekinumab Then Ustekinumab
Number analyzed (Participants) | 8 | 6 | 3 | 4
Participants | 6 | 5 | 1 | 2

3. Secondary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (SAEs)
Description: SAE is any untoward medical occurrence that at any dose may results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product. Treatment-emergent SAEs were defined as SAEs with onset or worsening on or after date of first dose of study intervention through the day of last dose.
Time Frame: Double-blind period: Double-blind Week 0 up to end of double-blind treatment period (56.1 weeks); OLE: OL Week 0 up to end of OLE treatment period (48.1 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Double-blind: Placebo: In double-blind period, participants received body weight-range placebo intravenous (IV) infusion at Week 0 followed by placebo subcutaneous (SC) injection administration, 8 weeks after the initial IV dose, then every 8 weeks (q8w) thereafter until developing relapse or end of double-blind period, with starting the protocol defined oral GC taper regimen from Week 2. Participants who received placebo in double-blind period and reached oral GC dose of 5 mg/day or less were terminated from study intervention administration and underwent early-term visit after completion of double-blind period.
Arm/Group | Double-blind: Placebo | Double-blind: Ustekinumab | OLE: Placebo Then Ustekinumab | OLE: Ustekinumab Then Ustekinumab
Number analyzed (Participants) | 8 | 6 | 3 | 4
Participants | 1 | 1 | 0 | 1

4. Secondary Outcome: Time to Relapse of TAK According to Kerr's Criteria Through the End of Double-blind Period
Description: ToR was defined from the date of randomization to the judged date of relapse through the EDBP based on Kerr's definition: participants who met 2 or more categories in the following 4 categories were considered as relapse: systemic (objective):body temperature >=38.0°C, weight loss >2kg in 4 weeks, arthralgia, swelling & tenderness =>2 joints; systemic (subjective):malaise, myalgia, headache, dizziness/vertigo at >= grade 2, high inflammation markers (C-reactive protein >=1.0mg/dL, erythrocyte sedimentation rate >=30mm/hr), vascular symptoms:renovascular hypertension: if normal BP <120/80mmHg risen to >=140/90mmHg, or if normal BP >=120/80mmHg, diastolic BP risen by >=20mmHg, new bruits/loss of pulse/difference in systolic BP between left and right by >=10mmHg/tenderness/spontaneous pain in carotid artery/chest/back region, aortic valve incompetence; ischemic symptoms:abdominal pain, seizure, syncope, intermittent claudication, ischemic cardiac pain.
Time Frame: From double-blind Week 0 up to end of double-blind period (up to 71.1 weeks)
Population: FAS includes all randomized participants who received at least 1 dose of study intervention through double-blind period.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Double-blind: Placebo | Double-blind: Ustekinumab
Number analyzed (Participants) | 8 | 6
Weeks | 12.64 [12.14 to NA] — Upper limit of 95% CI was not estimable due to less number of participants with events due to early study termination. | 11.14 [4.14 to NA] — Upper limit of 95% CI was not estimable due to less number of participants with events due to early study termination.

5. Secondary Outcome: Time to Relapse of TAK Based on Clinical Symptoms Through the End of Double-blind Period
Description: Time (in weeks) to relapse of TAK: time from randomization to the 1st relapse through the EDBP according to protocol-defined criteria with 5 categories: systemic (objective):body temperature >=38.0°C, weight loss >2kg in 4 weeks, arthralgia, swelling and tenderness =>2 joints; systemic (subjective):malaise, myalgia, headache, dizziness/vertigo at >= grade 2, high inflammation markers (C-reactive protein >=1.0mg/dL, erythrocyte sedimentation rate >=30mm/hr), vascular symptoms:renovascular hypertension: if normal BP <120/80mmHg risen to >=140/90mmHg, or if normal BP >=120/80mmHg, diastolic BP risen by >=20mmHg, new bruits/loss of pulse/difference in systolic BP between left and right by >=10mmHg/tenderness/spontaneous pain in carotid artery/chest/back region, aortic valve incompetence; ischemic symptoms:abdominal pain, seizure, syncope, intermittent claudication, ischemic cardiac pain. Time to relapse was calculated by each category independently. Relapse:>=2 categories met criteria.
Time Frame: From double-blind Week 0 up to end of double-blind period (up to 71.1 weeks)
Population: FAS included all randomized participants who received at least 1 dose of study intervention through double-blind period.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Double-blind: Placebo | Double-blind: Ustekinumab
Number analyzed (Participants) | 8 | 6
weeks | 12.14 [2.14 to NA] — Upper limit of 95% CI was not estimable due to less number of participants with events due to early study termination. | 4.14 [2.14 to NA] — Upper limit of 95% CI was not estimable due to less number of participants with events due to early study termination.

6. Secondary Outcome: Time to Relapse of TAK in Each of the 5 Categories (Within Protocol-defined Criteria) Through the End of Double-blind Period
Description: Time to relapse of TAK: time from randomization date to the 1st relapse through the EDBP according to protocol-defined criteria with 5 categories: systemic (objective):body temperature >=38.0°C, weight loss >2kg in 4 weeks, arthralgia, swelling and tenderness =>2 joints; systemic (subjective):malaise, myalgia, headache, dizziness/vertigo at >= grade 2, high inflammation markers (C-reactive protein >=1.0mg/dL, erythrocyte sedimentation rate >=30mm/hr), vascular symptoms:renovascular hypertension: if normal BP <120/80mmHg risen to >=140/90mmHg, or if normal BP >=120/80mmHg, diastolic BP risen by >=20mmHg, new bruits/loss of pulse/difference in systolic BP between left and right by >=10mmHg/tenderness/spontaneous pain in carotid artery/chest/back region, aortic valve incompetence; ischemic symptoms:abdominal pain, seizure, syncope, intermittent claudication, ischemic cardiac pain. Time to relapse was calculated by each category independently. Relapse:>=2 categories met criteria.
Time Frame: From double-blind Week 0 up to end of double-blind period (up to 71.1 weeks)
Population: FAS includes all randomized participants who received at least 1 dose of study intervention through double-blind period. Here, '0' in the number analyzed field signifies that no participants were in relapse.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Double-blind: Placebo | Double-blind: Ustekinumab
Number analyzed (Participants) | 8 | 6
weeks
  Systemic Symptoms (Objective Assessment) | 14.00 [12.14 to NA] — NA indicates that lower limit of CI was not estimable due to insufficient number of participants with events at study closure. | NA [12.14 to NA] — NA indicates that median and lower limit of CI were not estimable due to insufficient number of participants with events at study closure.
  Systemic Symptoms (Subjective Assessment) | 12.64 [12.14 to NA] — NA indicates that lower limit of CI was not estimable due to insufficient number of participants with events at study closure. | 10.00 [2.14 to NA] — NA indicates that lower limit of CI was not estimable due to insufficient number of participants with events at study closure.
  Elevated Inflammation Markers | 13.14 [8.14 to NA] — NA indicates that lower limit of CI was not estimable due to insufficient number of participants with events at study closure. | 12.14 [4.14 to NA] — NA indicates that lower limit of CI was not estimable due to insufficient number of participants with events at study closure.
  Vascular Signs And Symptoms | 12.14 [2.14 to NA] — NA indicates that lower limit of CI was not estimable due to insufficient number of participants with events at study closure. | 7.14 [2.14 to NA] — NA indicates that lower limit of CI was not estimable due to insufficient number of participants with events at study closure.
  Ischemic Symptoms: number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Participants With Relapse of TAK in Each of the 5 Categories (Within Protocol-defined Criteria) Through the End of Double-blind Period
Description: Percentage of participants with time to relapse of TAK through the EDBP were reported. Protocol-defined criteria consisted of 5 categories: systemic (objective):body temperature >=38.0°C, weight loss >2kg in 4 weeks, arthralgia, swelling & tenderness =>2 joints; systemic (subjective):malaise, myalgia, headache, dizziness/vertigo at >= grade 2, high inflammation markers (C-reactive protein >=1.0mg/dL, erythrocyte sedimentation rate >=30mm/hr), vascular symptoms:renovascular hypertension: if normal BP <120/80mmHg risen to >=140/90mmHg, or if normal BP >=120/80mmHg, diastolic BP risen by >=20mmHg, new bruits/loss of pulse/difference in systolic BP between left and right by >=10mmHg/tenderness/spontaneous pain in carotid artery/chest/back region, aortic valve incompetence; ischemic symptoms: abdominal pain, seizure, syncope, intermittent claudication, ischemic cardiac pain.
Time Frame: From double-blind Week 0 up to end of double-blind period (up to 71.1 weeks)
Population: FAS includes all randomized participants who received at least 1 dose of study intervention through double-blind period.
Measure: Number; unit: percentage of participants
Arm/Group | Double-blind: Placebo | Double-blind: Ustekinumab
Number analyzed (Participants) | 8 | 6
percentage of participants
  Systemic Symptoms (Objective Assessment) | 25.0 | 16.7
  Systemic Symptoms (Subjective Assessment) | 37.5 | 50.0
  Elevated Inflammation Markers | 50.0 | 50.0
  Vascular Signs And Symptoms | 50.0 | 100.0
  Ischemic Symptoms | 0 | 0

8. Secondary Outcome: Cumulative Oral Glucocorticoid (GC) Dose Through the End of Double-blind Period
Description: Cumulative oral GC dose (prednisolone or equivalent) through the end of double-blind period were reported. If the participant had relapse, oral GC dose (prednisolone or equivalent) used from randomization date to last observed date prior to the date of relapse were included in the analysis and if the participant had no relapse then oral GC dose used from randomization to last observed date through the end of double-blind period were included in the analysis.
Time Frame: From double-blind Week 0 up to end of double-blind period (up to 71.1 weeks)
Population: FAS includes all randomized participants who received at least 1 dose of study intervention through double-blind period.
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | Double-blind: Placebo | Double-blind: Ustekinumab
Number analyzed (Participants) | 8 | 6
milligrams (mg) | 1043.6 (367.27) | 1319.1 (697.67)

9. Secondary Outcome: Change From Baseline in Oral GC Dose Through the End of Double-blind Period
Description: Change from baseline in oral GC dose through the end of double-blind period were reported. Change from baseline was defined as the change between the GC dose at randomization and the last observed GC dose. If the participant had relapse, oral GC dose (prednisolone or equivalent) used from randomization date to last observed date prior to the date of relapse were included in the analysis and if the participant had no relapse then oral GC dose used from randomization to last observed date through the end of double-blind period were included in the analysis.
Time Frame: Baseline (double-blind Week 0) up to end of double-blind period (up to 71.1 weeks)
Population: FAS includes all randomized participants who received at least 1 dose of study intervention through double-blind period.
Measure: Mean (Standard Deviation); unit: milligrams per day (mg/day)
Arm/Group | Double-blind: Placebo | Double-blind: Ustekinumab
Number analyzed (Participants) | 8 | 6
milligrams per day (mg/day) | -11.3 (3.73) | -12.1 (6.25)

10. Secondary Outcome: Number of Participants Achieving GC Dose of 5 mg/Day or Less Through the End of Double-blind Period
Description: Number of participants who achieved GC dose of 5 mg/day or less through the end of double-blind period were reported.
Time Frame: From double-blind Week 0 up to end of double-blind period (up to 71.1 weeks)
Population: FAS includes all randomized participants who received at least 1 dose of study intervention through double-blind period.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind: Placebo | Double-blind: Ustekinumab
Number analyzed (Participants) | 8 | 6
Participants | 3 | 1

11. Secondary Outcome: Change From Baseline in Imaging Evaluation of Vessel Involvement (Average Percentage of Dilation) at the End of Double-blind Period
Description: Change from baseline in average percentage of dilation for abnormal vessel segments through the end of double-blind period was reported. Assessment was performed using computed tomography angiography (CTA) or magnetic resonance angiography (MRA). For a participant, the time point at which the 1st relapse developed or discontinuation from double-blind period was considered as the end of double-blind period.
Time Frame: Baseline (double-blind Week 0) and double-blind relapse (up to 14 weeks for Placebo arm; up to 48 weeks for ustekinumab arm)
Population: FAS includes all randomized participants who received at least 1 dose of study intervention through double-blind period. Here, '0' in the number of participants analyzed field of arm 'Double-blind: Placebo' signifies that no participants were available for analysis because placebo group did not have abnormal dilation at double-blind relapse visit. Here, 'N' (number of participants analyzed): who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of Dilation
Arm/Group | Double-blind: Placebo | Double-blind: Ustekinumab
Number analyzed (Participants) | 0 | 2
Percentage of Dilation |  | -3.95 (5.586)

12. Secondary Outcome: Change From Baseline in Imaging Evaluation of Vessel Involvement (Average Percentage of Stenosis) Through the End of Double-blind Period
Description: Change from baseline in average percentage of stenosis for abnormal vessel segments through the end of double-blind period was reported. Assessment was performed using CTA or MRA. For a participant, the time point at which the 1st relapse developed or discontinuation from double-blind period was considered as the end of double-blind period.
Time Frame: Baseline (double-blind Week 0), Week 24, Week 48, and double-blind relapse (up to 14 weeks for Placebo arm; up to 48 weeks for ustekinumab arm)
Population: FAS: who received at least 1 dose of study intervention through double-blind period. Here, '0' in the number analyzed field of 'Double-blind: Placebo' arm signifies that no participant was available for analysis because all placebo group participants either relapsed or discontinued the study before Week 24. Here, 'N' (number of participants analyzed): who were evaluable for this outcome measure and 'n' (number analysed): number of participants analyzed at each specified timepoints.
Measure: Mean (Standard Deviation); unit: Percentage of Stenosis
Arm/Group | Double-blind: Placebo | Double-blind: Ustekinumab
Number analyzed (Participants) | 2 | 4
Percentage of Stenosis
  Double-blind Week 24: number analyzed (Participants) | 0 | 1
  Double-blind Week 24 |  | -11.39 (NA) — Standard deviation was not estimable for 1 participant.
  Double-blind Week 48: number analyzed (Participants) | 0 | 1
  Double-blind Week 48 |  | -12.62 (NA) — Standard deviation was not estimable for 1 participant.
  Double-blind Relapse | -7.15 (10.105) | -13.94 (22.24)

13. Secondary Outcome: Change From Baseline in Imaging Evaluation of Average Arterial Wall Thickness Through the End of Double-blind Period
Description: Change from baseline in average wall thickness for abnormal segments through the end of double-blind period was reported. Assessment was performed using CTA or MRA. For a participant, the time point at which the 1st relapse developed or discontinuation from double-blind period was considered as the end of double-blind period.
Time Frame: as for outcome 12
Population: FAS: who received at least 1 dose of study intervention through double-blind period. Here, '0' in the number analyzed field of 'Double-blind: Placebo' arm signifies that no participant was available for analysis because all placebo group participants either relapsed or discontinued the study before Week 24. Here, 'N' (number of participants analyzed): who were evaluable for this outcome measure and 'n' (number analyzed):number of participants analyzed at each specified timepoints.
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- Double-blind : Placebo: In double-blind period, participants received body weight-range placebo intravenous (IV) infusion at Week 0 followed by placebo subcutaneous (SC) injection administration, 8 weeks after the initial IV dose, then every 8 weeks (q8w) thereafter until developing relapse or end of double-blind period, with starting the protocol defined oral GC taper regimen from Week 2. Participants who received placebo in double-blind period and reached oral GC dose of 5 mg/day or less were terminated from study intervention administration and underwent early-term visit after completion of double-blind period.
Arm/Group | Double-blind : Placebo | Double-blind: Ustekinumab
Number analyzed (Participants) | 1 | 1
millimeters
  Double-blind Week 24: number analyzed (Participants) | 0 | 1
  Double-blind Week 24 |  | -1.25 (NA) — Standard deviation was not estimable for 1 participant.
  Double-blind Week 48: number analyzed (Participants) | 0 | 1
  Double-blind Week 48 |  | -1.25 (NA) — Standard deviation was not estimable for 1 participant.
  Double-blind Relapse | -1.00 (NA) — Standard deviation was not estimable for 1 participant. | 1.00 (NA) — Standard deviation was not estimable for 1 participant.

14. Secondary Outcome: Imaging Evaluation: Number of Participants With Mural Contrast Enhancement Through the End of Double-blind Period
Description: Number of participants with mural contrast enhancement through the end of double-blind period were reported. The mural contrast enhancement were assessed for imaging evaluation using CTA or MRA. For a participant, the time point at which the 1st relapse developed or discontinuation from double-blind period was considered as the end of double-blind period.
Time Frame: as for outcome 12
Population: FAS: who received at least 1 dose of study intervention through double-blind period. Here, '0' in the number analyzed field of Double-blind: Placebo arm signifies that no participant was available for analysis because all placebo group participants either relapsed or discontinued the study before Week 24. Here, 'N' (number of participants analyzed): who were evaluable for this outcome measure and 'n' (number analyzed): number of participants analyzed at each specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind: Placebo | Double-blind: Ustekinumab
Number analyzed (Participants) | 7 | 6
Participants
  Baseline (Week 0) | 1 | 1
  Double-blind Week 24: number analyzed (Participants) | 0 | 1
  Double-blind Week 24 |  | 1
  Double-blind Week 48: number analyzed (Participants) | 0 | 1
  Double-blind Week 48 |  | 1
  Double-blind Relapse: number analyzed (Participants) | 4 | 4
  Double-blind Relapse | 0 | 1

15. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP) Through the End of Double-blind Period
Description: Change from baseline in CRP (as inflammatory marker) through the end of double-blind period were reported. For a participant, the time point at which the 1st relapse developed or discontinuation from double-blind period was considered as the end of double-blind period.
Time Frame: Baseline (double-blind Week 0), Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, and double-blind relapse (up to 14 weeks for Placebo arm; up to 48 weeks for ustekinumab arm)
Population: FAS includes all randomized participants who received at least 1 dose of study intervention through double-blind period. Here, '0' in the number analyzed field of arm 'Double-blind: Placebo', signifies that no participant was available for analysis because all placebo group participants either relapsed or discontinued the study before Week 24. Here, 'n' (number analyzed) signifies number of participants analyzed at each specified timepoints.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Double-blind: Placebo | Double-blind: Ustekinumab
Number analyzed (Participants) | 8 | 6
milligrams per deciliter (mg/dL)
  Double-blind Week 2: number analyzed (Participants) | 8 | 5
  Double-blind Week 2 | -0.003 (0.0539) | 0.558 (0.9585)
  Double-blind Week 4 | 0.529 (1.4639) | 0.858 (1.6216)
  Double-blind Week 8: number analyzed (Participants) | 6 | 4
  Double-blind Week 8 | 0.918 (1.3851) | 0.333 (0.3505)
  Double-blind Week 12: number analyzed (Participants) | 4 | 3
  Double-blind Week 12 | 1.475 (0.5132) | 1.170 (1.0333)
  Double-blind Week 16: number analyzed (Participants) | 0 | 1
  Double-blind Week 16 |  | -0.010 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Week 20: number analyzed (Participants) | 0 | 1
  Double-blind Week 20 |  | -0.030 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Week 24: number analyzed (Participants) | 0 | 1
  Double-blind Week 24 |  | 0.00 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Week 28: number analyzed (Participants) | 0 | 1
  Double-blind Week 28 |  | 0.00 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Week 32: number analyzed (Participants) | 0 | 1
  Double-blind Week 32 |  | 0.310 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Week 36: number analyzed (Participants) | 0 | 1
  Double-blind Week 36 |  | 0.060 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Week 40: number analyzed (Participants) | 0 | 1
  Double-blind Week 40 |  | -0.020 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Week 44: number analyzed (Participants) | 0 | 1
  Double-blind Week 44 |  | 0.300 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Week 48: number analyzed (Participants) | 0 | 1
  Double-blind Week 48 |  | -0.010 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Week 52: number analyzed (Participants) | 0 | 1
  Double-blind Week 52 |  | 0.010 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Week 56: number analyzed (Participants) | 0 | 1
  Double-blind Week 56 |  | 0.130 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Relapse: number analyzed (Participants) | 4 | 4
  Double-blind Relapse | 2.043 (1.5661) | 2.598 (3.2988)

16. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) Through the End of Double-blind Period
Description: Change from baseline in ESR (as inflammatory marker) through the end of double-blind period were reported. For a participant, the time point at which the 1st relapse developed or discontinuation from double-blind period was considered as the end of double-blind period.
Time Frame: as for outcome 15
Population: FAS includes all randomized participants who received at least 1 dose of study intervention through double-blind period. Here, '0' in the number analyzed field of "Double-blind: Placebo" arm signifies that no participant was available for analysis because all placebo group participants either relapsed or discontinued the study before Week 24. Here, 'n' (number analyzed) signifies number of participants analyzed at each specified timepoints.
Measure: Mean (Standard Deviation); unit: millimeters per hour (mm/h)
Arm/Group | Double-blind: Placebo | Double-blind: Ustekinumab
Number analyzed (Participants) | 8 | 6
millimeters per hour (mm/h)
  Double-blind Week 2: number analyzed (Participants) | 8 | 5
  Double-blind Week 2 | 0.13 (1.246) | 1.20 (8.349)
  Double-blind Week 4 | 4.75 (11.841) | 4.33 (17.397)
  Double-blind Week 8: number analyzed (Participants) | 6 | 4
  Double-blind Week 8 | 6.67 (4.131) | 5.13 (7.028)
  Double-blind Week 12: number analyzed (Participants) | 4 | 3
  Double-blind Week 12 | 24.25 (15.174) | 15.50 (15.174)
  Double-blind Week 16: number analyzed (Participants) | 0 | 1
  Double-blind Week 16 |  | 1.00 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Week 20: number analyzed (Participants) | 0 | 1
  Double-blind Week 20 |  | -2.00 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Week 24: number analyzed (Participants) | 0 | 1
  Double-blind Week 24 |  | -2.00 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Week 28: number analyzed (Participants) | 0 | 1
  Double-blind Week 28 |  | 12.00 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Week 32: number analyzed (Participants) | 0 | 1
  Double-blind Week 32 |  | 13.00 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Week 36: number analyzed (Participants) | 0 | 1
  Double-blind Week 36 |  | 2.00 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Week 40: number analyzed (Participants) | 0 | 1
  Double-blind Week 40 |  | 2.00 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Week 44: number analyzed (Participants) | 0 | 1
  Double-blind Week 44 |  | 0.00 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Week 48: number analyzed (Participants) | 0 | 1
  Double-blind Week 48 |  | -2.00 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Week 52: number analyzed (Participants) | 0 | 1
  Double-blind Week 52 |  | -2.00 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Week 56: number analyzed (Participants) | 0 | 1
  Double-blind Week 56 |  | 20.00 (NA) — Stand deviation was not estimable for 1 participant.
  Double-blind Relapse: number analyzed (Participants) | 4 | 4
  Double-blind Relapse | 28.25 (15.500) | 18.63 (9.741)

17. Secondary Outcome: Serum Concentrations of Ustekinumab in Participants Receiving Ustekinumab During Double-blind Phase
Description: Serum concentrations of ustekinumab was reported during double-blind Phase. For a participant, the time point at which the 1st relapse developed or discontinuation from double-blind period was considered as the end of double-blind period.
Time Frame: Pre-dose (double-blind Week 0), Post-dose: Week 0, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, double-blind relapse (up to 48 weeks)
Population: The pharmacokinetic (PK) analysis set was defined as participants who received at least 1 complete dose of ustekinumab and had at least 1 valid postdose PK data. Here, 'n' (number analyzed) signifies number of participants analyzed at each specified timepoints. For this outcome measure, as pre-planned, data collection and analysis was not performed for the placebo arm.
Measure: Mean (Standard Deviation); unit: micrograms per millilitres (mcg/mL)
Arm/Group | Double-blind: Ustekinumab
Number analyzed (Participants) | 6
micrograms per millilitres (mcg/mL)
  Pre-dose (Week 0) | NA (NA) — Here, 'NA' signifies that mean and standard deviation could not be estimated as the analyzed values were below the lower limit of quantification (LLOQ) (0.1688 mcg/mL).
  Post-dose (Week 0) | 135.644 (33.2099)
  Week 2: number analyzed (Participants) | 5
  Week 2 | 40.470 (8.5492)
  Week 4 | 21.630 (3.5437)
  Week 8: number analyzed (Participants) | 5
  Week 8 | 8.663 (2.9795)
  Week 12: number analyzed (Participants) | 3
  Week 12 | 7.762 (0.7537)
  Week 16: number analyzed (Participants) | 1
  Week 16 | 3.811 (NA) — Standard deviation was not evaluable for 1 participant.
  Week 20: number analyzed (Participants) | 1
  Week 20 | 4.970 (NA) — Standard deviation was not evaluable for 1 participant.
  Week 24: number analyzed (Participants) | 1
  Week 24 | 2.195 (NA) — Standard deviation was not evaluable for single participant.
  Week 28: number analyzed (Participants) | 1
  Week 28 | 5.323 (NA) — Standard deviation was not evaluable for 1 participant.
  Week 32: number analyzed (Participants) | 1
  Week 32 | 2.033 (NA) — Standard deviation was not evaluable for 1 participant.
  Week 36: number analyzed (Participants) | 1
  Week 36 | 3.984 (NA) — Standard deviation was not evaluable for 1 participant.
  Week 40: number analyzed (Participants) | 1
  Week 40 | 1.695 (NA) — Standard deviation was not evaluable for 1 participant.
  Week 44: number analyzed (Participants) | 1
  Week 44 | 4.958 (NA) — Standard deviation was not evaluable for 1 participant.
  Week 48: number analyzed (Participants) | 1
  Week 48 | 2.121 (NA) — Standard deviation was not evaluable for 1 participant.
  Week 52: number analyzed (Participants) | 1
  Week 52 | 6.447 (NA) — Standard deviation was not evaluable for 1 participant.
  Week 56: number analyzed (Participants) | 1
  Week 56 | 2.596 (NA) — Standard deviation was not evaluable for 1 participant.
  Week 60: number analyzed (Participants) | 1
  Week 60 | 3.244 (NA) — Standard deviation was not evaluable for 1 participant.
  Double-blind: Relapse: number analyzed (Participants) | 2
  Double-blind: Relapse | 13.437 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as the analyzed value was below the LLOQ (0.1688 mcg/mL).

18. Secondary Outcome: Serum Concentrations of Ustekinumab in Participants Receiving Ustekinumab During Open-label Extension Phase
Description: Serum concentrations of ustekinumab was reported during OLE Phase.
Time Frame: Pre-dose (OL Week 0), Post-dose: OL Week 0, OL Weeks 8, 16, 24, 32, 40, 48, 52, and 56
Population: PK analysis set: who experienced relapse in double-blind period and received at least 1 complete dose of ustekinumab and had at least 1 valid postdose PK data from OL Week 0 to end of OLE period. Here, '0' in the number analyzed field of second arm signifies that no participant was available for analysis because all participants were relapsed before OL Week 48. Here, 'n' (number analyzed): number of participants analyzed at each specified timepoints.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | OLE: Placebo Then Ustekinumab | OLE: Ustekinumab Then Ustekinumab
Number analyzed (Participants) | 3 | 4
mcg/mL
  Pre-dose OL Week 0 | NA (NA) — Here, 'NA' signifies that mean and standard deviation could not be estimated as the analyzed value was below the LLOQ (0.1688 mcg/mL). | 4.765 (2.1977)
  Post-dose OL Week 0 | 126.394 (15.5782) | 132.580 (36.2574)
  OL Week 8: number analyzed (Participants) | 3 | 3
  OL Week 8 | 15.830 (7.3113) | 10.912 (4.5891)
  OL Week 16: number analyzed (Participants) | 2 | 2
  OL Week 16 | 7.253 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as the analyzed value was below the LLOQ (0.1688 mcg/mL). | 7.560 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as the analyzed value was below the LLOQ (0.1688 mcg/mL).
  OL Week 24: number analyzed (Participants) | 3 | 1
  OL Week 24 | 8.844 (4.3775) | 4.807 (NA) — Standard deviation was not evaluable for 1 participant.
  OL Week 32: number analyzed (Participants) | 2 | 1
  OL Week 32 | 6.096 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as the analyzed value was below the LLOQ (0.1688 mcg/mL). | 3.870 (NA) — Standard deviation was not evaluable for 1 participant.
  OL Week 40: number analyzed (Participants) | 1 | 1
  OL Week 40 | 3.911 (NA) — Standard deviation was not evaluable for 1 participant. | 3.911 (NA) — Standard deviation was not evaluable for 1 participant.
  OL Week 48: number analyzed (Participants) | 1 | 0
  OL Week 48 | 3.719 (NA) — Standard deviation was not evaluable for 1 participant. |
  OL Week 52: number analyzed (Participants) | 1 | 0
  OL Week 52 | 9.676 (NA) — Standard deviation was not evaluable for 1 participant. |
  OL Week 56: number analyzed (Participants) | 1 | 0
  OL Week 56 | 3.710 (NA) — Standard deviation was not evaluable for 1 participant. |

19. Secondary Outcome: Number of Participants With Positive Anti-ustekinumab Antibodies Through End of Double-blind Period
Description: Number of participants with positive anti-ustekinumab antibodies were reported.
Time Frame: From double-blind Week 0 up to end of double-blind period (up to 71.1 weeks)
Population: The immunogenicity analysis set was defined as all participants who received at least 1 dose of ustekinumab and had at least 1 postdose valid immunogenicity data. For this outcome measure, as pre-planned, data collection and analysis was not performed for the placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind: Ustekinumab
Number analyzed (Participants) | 6
Participants | 0

20. Secondary Outcome: Number of Participants With Positive Anti-ustekinumab Antibodies Through End of OLE Period
Description: Number of participants with positive anti-ustekinumab antibodies were reported.
Time Frame: From OL Week 0 up to end of OLE period (up to 63.1 weeks)
Population: The immunogenicity analysis set was defined as all participants who received at least 1 dose of ustekinumab and had at least 1 postdose valid immunogenicity data. In ustekinumab arm N included all participants who were initially randomized to ustekinumab arm.
Measure: Count of Participants; unit: Participants
Arm/Group | OLE: Placebo Then Ustekinumab | OLE: Ustekinumab Then Ustekinumab
Number analyzed (Participants) | 3 | 6
Participants | 0 | 0

21. Secondary Outcome: Number of Participants With TEAEs by System Organ Class (SOC) With a Frequency Threshold of 5 Percent (%) or More
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with the study intervention. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study intervention through the day of last dose. If same participant had more than one AE within the same SOC, that participant is counted only once in the below data table.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind: Placebo | Double-blind: Ustekinumab | OLE: Placebo Then Ustekinumab | OLE: Ustekinumab Then Ustekinumab
Number analyzed (Participants) | 8 | 6 | 3 | 4
Participants
  Ear and Labyrinth Disorders | 0 | 1 | 0 | 0
  Eye Disorders | 2 | 2 | 0 | 0
  Gastrointestinal Disorders | 3 | 0 | 1 | 2
  General Disorders and Administration Site Conditions | 0 | 4 | 0 | 2
  Infections and Infestations | 1 | 6 | 0 | 0
  Injury, Poisoning and Procedural Complications | 1 | 3 | 1 | 1
  Investigations | 0 | 1 | 0 | 1
  Metabolism and Nutrition Disorders | 0 | 1 | 0 | 0
  Musculoskeletal and Connective Tissue Disorders | 1 | 1 | 0 | 0
  Nervous System Disorders | 0 | 5 | 1 | 1
  Respiratory, Thoracic and Mediastinal Disorders | 0 | 0 | 0 | 2
  Skin and Subcutaneous Tissue Disorders | 4 | 0 | 0 | 0
  Vascular Disorders | 1 | 2 | 0 | 1

ADVERSE EVENTS:
Time Frame: Double-blind period: From double-blind Week 0 up to end of double-blind period (up to 71.1 weeks); OLE period: From OL-Week 0 up to end of OLE period (up to 63.1 weeks)
Description: Safety assessments were based on the safety analysis set included all participants who received at least 1 dose of study intervention through double-blind period and OLE period.
Groups:
- Double Blind: Placebo: In double-blind period, participants received placebo matched to ustekinumab as intravenous (IV) infusion at Week 0 followed by placebo subcutaneous (SC) injection administration, 8 weeks after the initial IV dose, then every 8 weeks (q8w) thereafter until developing relapse or end of double-blind period, with starting the protocol defined oral GC taper regimen from Week 2. Participants who received placebo in double-blind period and reached oral GC dose of 5 mg/day or less were terminated from study intervention administration and underwent early-term visit after completion of double-blind period.
- OLE Period: Placebo Then Ustekinumab: Participants who had relapse during the double-blind period, received rescue medication of >=doubled oral GC dose. These participants were assessed whether they achieved remission at the next scheduled dose administration visit (OL Week 0) from the relapse to enter OLE period and received ustekinumab 90 mg IV infusion at OL Week 0 followed by ustekinumab 90 mg SC injection at OL Week 8 and thereafter q8w in OLE period (maximum exposure: 48.1 weeks). Rest of the participants entered OLE period after end of double blind period and then they received ustekinumab 90 mg SC injection (maintenance dosing) q8w from OL Week 0 (maximum exposure: 48.1 weeks). Participants who received placebo (up to 8.1 weeks) in double-blind period received ustekinumab 90 mg SC injection (maintenance dosing) q8w from OL Week 0 till end of OLE period (maximum exposure: 48.1 weeks).
- OLE Period: Ustekinumab Then Ustekinumab: Participants who had relapse during the double-blind period, received rescue medication of >=doubled oral GC dose. These participants were assessed whether they achieved remission at the next scheduled dose administration visit (OL Week 0) from the relapse to enter OLE period and then they received ustekinumab 90 mg IV infusion at OL Week 0 followed by ustekinumab 90 mg SC injection at OL Week 8 and thereafter q8w till end of OLE period (maximum exposure: 48.1 weeks). Participants with no remission status received ustekinumab IV infusion at OL Week 0 and thereafter q8w till end of OLE period (maximum exposure 48.1 weeks). Rest of the participants entered OLE period after end of double-blind period and received ustekinumab 90 mg SC injection (maintenance dosing) q8w from OL Week 0 (maximum exposure: 48.1 weeks).
Arm/Group | Double Blind: Placebo | Double-blind: Ustekinumab | OLE Period: Placebo Then Ustekinumab | OLE Period: Ustekinumab Then Ustekinumab
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/6 | 0/3 | 1/4
Other Adverse Events (participants affected / at risk) | 6/8 | 5/6 | 1/3 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind: Placebo (N=8) | Double-blind: Ustekinumab (N=6) | OLE Period: Placebo Then Ustekinumab (N=3) | OLE Period: Ustekinumab Then Ustekinumab (N=4)
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Vascular Graft Infection (Infections and infestations) | 0 | 0 | 0 | 1
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Brachiocephalic Artery Stenosis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind: Placebo (N=8) | Double-blind: Ustekinumab (N=6) | OLE Period: Placebo Then Ustekinumab (N=3) | OLE Period: Ustekinumab Then Ustekinumab (N=4)
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Conjunctival Haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Posterior Capsule Opacification (Eye disorders) | 0 | 1 | 0 | 0
Retinal Vascular Disorder (Eye disorders) | 0 | 1 | 0 | 0
Visual Impairment (Eye disorders) | 1 | 0 | 0 | 0
Coating in Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dental Caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 2 | 0 | 1
Vaccination Site Pain (General disorders) | 0 | 2 | 0 | 0
Aspergillus Infection (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 1 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Tinea Pedis (Infections and infestations) | 0 | 1 | 0 | 0
Chillblains (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Postoperative Hypertension (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound Complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Sars-Cov-2 Test Positive (Investigations) | 0 | 0 | 0 | 1
Weight Decreased (Investigations) | 0 | 1 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Lacunar Infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Paralysis Recurrent Laryngeal Nerve (Nervous system disorders) | 0 | 0 | 0 | 1
Post Herpetic Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hand Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Takayasu's Arteritis (Vascular disorders) | 1 | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early by the sponsor due to difficulties in participant recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT04882072/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT04882072/SAP_001.pdf